CLINICAL TRIAL: NCT01520116
Title: A Phase 1/2a Randomized, Investigator-masked, Placebo- and Active-controlled, Dose-ranging Study of the Safety and Efficacy of ATS907 in Subjects With Primary Open Angle Glaucoma (POAG) and Ocular Hypertension
Brief Title: Study of the Safety and Efficacy of ATS907 in Subjects With Primary Open Angle Glaucoma (POAG) and Ocular Hypertension
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Altheos, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATS907-201
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Timolol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Stage 1 - Arm 1 - Dose 1 (Experimental)
  Interventions: Drug: Stage 1 - ATS907 - Dose 1
- Stage 1 - Arm 2 - Dose 2 (Experimental)
  Interventions: Drug: Stage 1 - ATS907 - Dose 2
- Stage 1 - Arm 3 - Dose 3 (Experimental)
  Interventions: Drug: Stage 1 - ATS907 - Dose 3
- Stage 1 - Arm 4 - Dose 4 (Experimental)
  Interventions: Drug: Stage 1 - ATS907 - Dose 4
- Stage 1 - Arm 5 - Vehicle (Placebo Comparator)
  Interventions: Drug: Stage 1 - Vehicle
- Stage 2 - Arm 1 - Dose A - to be selected based on Stage 1 (Experimental)
  Interventions: Drug: Stage 2 - ATS907 - Dose A - to be selected based on Stage 1
- Stage 2 - Arm 2 - Dose B - to be selected based on Stage 1 (Experimental)
  Interventions: Drug: Stage 2 - ATS907 - Dose B - to be selected based on Stage 1
- Stage 2 - Arm 3 -Timoptic 0.5% BID (Active Comparator)
  Interventions: Drug: Timoptic

INTERVENTIONS:
Drug: Stage 1 - ATS907 - Dose 1 — QD and/or BID dosing for 28 days
  Arms: Stage 1 - Arm 1 - Dose 1
Drug: Stage 1 - ATS907 - Dose 2 — QD and/or BID dosing for 28 days
  Arms: Stage 1 - Arm 2 - Dose 2
Drug: Stage 1 - ATS907 - Dose 3 — QD and/or BID dosing for 28 days
  Arms: Stage 1 - Arm 3 - Dose 3
Drug: Stage 1 - ATS907 - Dose 4 — QD and/or BID dosing for 28 days
  Arms: Stage 1 - Arm 4 - Dose 4
Drug: Stage 1 - Vehicle — QD and/or BID dosing for 28 days
  Arms: Stage 1 - Arm 5 - Vehicle
Drug: Stage 2 - ATS907 - Dose A - to be selected based on Stage 1 — QD and/or BID dosing for 4 days
  Arms: Stage 2 - Arm 1 - Dose A - to be selected based on Stage 1
Drug: Stage 2 - ATS907 - Dose B - to be selected based on Stage 1 — QD and/or BID dosing for 4 days
  Arms: Stage 2 - Arm 2 - Dose B - to be selected based on Stage 1
Drug: Timoptic — 0.5%
  Arms: Stage 2 - Arm 3 -Timoptic 0.5% BID

SUMMARY:
This randomized dose-ranging study will evaluate the safety, tolerability, and preliminary efficacy (reduction in intraocular pressure) of multiple dose levels of ATS907, vehicle, or latanoprost in subjects with primary open angle glaucoma or ocular hypertension. In the first portion, approximately 75 subjects will be randomized to receive either ATS907 or vehicle eye drops for up to 28 days, administered both once and twice daily. In the second portion, up to 180 subjects will be randomized to receive either ATS907 or latanoprost for up to 28 days. Plasma pharmacokinetics will also be evaluated during the first portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Diagnosis of open angle glaucoma (OAG) or ocular hypertension (OHT) in both eyes
* Unmedicated (post-washout) IOP ≥ 23 mm Hg at 2 eligibility visits: 07:00-09:00 hr on Days O and 1 and IOP > 18 mm Hg at 15:00-17:00 on Day 0 (Stage 1)
* Unmedicated (post-washout) IOP criteria after wash out < 32 mm Hg OU at all times points (Stage 1)
* Unmedicated (post-washout) IOP ≥ 24 mm Hg at 2 eligibility visits: 07:00-09:00 hr on Days O and 1 and IOP > 21 mm Hg at 9:00-17:00 on Day 0 (Stage 2)
* Unmedicated (post-washout) IOP criteria after wash out < 36 mm Hg OU at all times points (Stage 2)
* Corrected visual acuity in each eye +1.0 logMAR or better by ETDRS in each eye (equivalent to 20/200)
* Must be willing to discontinue the use of all ocular hypotensive medications in both eyes prior to and during the entire course of the study

Exclusion Criteria:

* Ophthalmic (in either eye)

  1. Glaucoma: pseudoexfoliation, steroid induced, pigment dispersion glaucoma, and or history of angle closure. Previous glaucoma intraocular surgery or glaucoma laser procedures in study eye(s). Prior laser glaucoma surgery is permitted in the non study eye
  2. Refractive surgery in study eye (e.g., radial keratotomy, PRK, LASIK, etc.)
  3. Cataract surgery and or other intraocular surgery within three months prior to Screening in either eye.
  4. History within 3 months prior to Screening of clinically significant moderate or severe chronic or active ocular infection, inflammation, blepharitis, dermatitis, uveitis or conjunctivitis.
  5. Clinically significant corneal dystrophy, epithelial and or endothelial disease, corneal irregularities and or scarring such that reliable applanation tonometry would prevented.
  6. Contact lens wear during the duration of the study.
  7. Clinically significant ocular disease (e.g. diabetic retinopathy, macular degeneration, or uveitis) which might interfere or progress during the study.
  8. Central corneal thickness < 480 or > 600 μm in the study eye
* Systemic

  1. Clinically significant abnormalities in laboratory tests at screening.
  2. Clinically significant systemic disease (e.g., uncontrolled diabetes, uncontrolled hyper or hypotension, hepatic, renal, endocrine or cardiovascular disorders). Participation in any investigational study within the past 30 days.
  3. Changes of systemic medication that could have a substantial effect on IOP and or systemic blood pressure within 7 days prior to Baseline (Day 0).
  4. Women of childbearing potential who are pregnant, nursing, planning a pregnancy, or not using a medically acceptable form of birth control. An adult woman is considered to be of childbearing potential unless she is one year post-menopausal or three months post-surgical sterilization. All females of childbearing potential must have a negative urine pregnancy test result at the Screening visit and a negative urine and serum pregnancy at Baseline (Day 0) and must not intend to become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Mean Change in Intraocular Pressure from Baseline | Stage 1: Days 14, 21 and 28; Stage 2: Day 4

SECONDARY OUTCOMES:
Observed Intraocular Pressure and % change from Baseline IOP | Stage 1: Days 0, 1, 4, 14, 21, 28; Stage 2: Days 0, 4
Mean observed, mean change from Baseline and mean % change from Baseline for the mean diurnal IOP | Stage 1: Days 0, 1, 4, 14, 21, 28; Stage 2: Days 0, 4

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Wirostko, MD, Study Chair — Altheos, Inc.
Locations (5):
- United States (5):
  - Artesia, California
  - Glendale, California
  - Saint Joseph, Michigan
  - Cleveland, Ohio
  - San Antonio, Texas